CLINICAL TRIAL: NCT06537791
Title: Multidisciplinary Home-Based Rehabilitation Program for Individuals With Disabilities: A Retrospective Study
Brief Title: Impact of Home-Based Rehabilitation on Motor Function and Mood in Individuals With Disabilities
Acronym: HB-Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0020
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Diseases; Neurological Diseases
Keywords: Musculoskeletal Disabilities; Neurological Disabilities; Berg Balance Scale; Beck Depression Inventory; Multidisciplinary Rehabilitation; Home-Based Care; Physical Rehabilitation; Mental Health Assessment; Fall Risk Reduction; Patient-Centered Care
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-Based Rehabilitation Program (Experimental): Participants in this arm will receive a multidisciplinary home-based rehabilitation program. The intervention includes 32 sessions of physical therapy, 8 sessions of occupational therapy, 4 sessions of nutrition counseling, 8 sessions of psychological support, and 4 sessions of nursing and podiatry care. Each session lasts 60 minutes, and the total duration of the intervention is approximately 4 months. The program aims to improve motor function, balance, and mood among individuals with moderate neuromusculoskeletal disabilities.
  Interventions: Behavioral: Home-Based Rehabilitation Program

INTERVENTIONS:
Behavioral: Home-Based Rehabilitation Program — Physical Therapy: 32 sessions, 60 minutes each Occupational Therapy: 8 sessions, 60 minutes each Nutrition Counseling: 4 sessions, 60 minutes each Psychological Support: 8 sessions, 60 minutes each Nursing and Podiatry Care: 4 sessions, 60 minutes each Total Duration: Approximately 4 months

SUMMARY:
This study aims to evaluate the impact of a multidisciplinary home-based rehabilitation program on motor function and mood in individuals with moderate neuromusculoskeletal disabilities. Participants will receive personalized treatment plans over four months, including sessions in physical therapy, occupational therapy, nutrition, psychology, nursing, and podiatry. The study will measure motor function using the Berg Balance Scale and mood using the Beck Depression Inventory. This program will be conducted in the Magallanes region of Chile, involving participants recruited from the National Disability Registry.

DETAILED DESCRIPTION:
This study is designed to assess the effectiveness of a comprehensive home-based rehabilitation program for individuals with moderate neuromusculoskeletal disabilities. The intervention will include a multidisciplinary approach, involving a team of healthcare professionals who will provide a range of services tailored to each participant's needs. The services will include 32 sessions of physical therapy, 8 sessions of occupational therapy, 4 sessions of nutrition counseling, 8 sessions of psychological support, and 4 sessions of nursing and podiatry care. The intervention will span four months, with a total of 82 hours of therapy per participant.

Participants will be evaluated at the beginning and end of the program using the Berg Balance Scale to measure motor function and the Beck Depression Inventory to assess mood. The study aims to demonstrat improvements in motor function and balance, with a reduction in fall risk, and to explore changes in depression levels among the participants.

Quality assurance procedures will include standardized training for all healthcare professionals involved, regular monitoring of therapy sessions, and adherence to established protocols for data collection and analysis. This study highlights the potential benefits of home-based rehabilitation programs and underscores the need for further research to explore long-term outcomes and additional measures to enhance patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with moderate neuromusculoskeletal disabilities.
* Participants referred by recognized medical institutions.
* Able to provide informed consent.

Exclusion Criteria:

* Individuals with severe cognitive impairments that hinder their ability to follow the rehabilitation program.
* Participants with acute medical conditions that require immediate hospitalization.
* Pregnant women.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Motor Function | From study start to the end of the intervention (4 months).
  Assessment of the improvement in motor function of the participants, measured using the Berg Balance Scale. This scale assesses balance through 14 common tasks performed in daily life. Scores range from 0 to 56 points, where 0 indicates a low level of balance and 56 indicates an excellent level of balance. A higher score on this scale represents a better outcome in terms of balance and motor function.

SECONDARY OUTCOMES:
Changes in Depression Levels | From study start to the end of the intervention (4 months).
  Assessment of changes in the participants' depression levels, measured using the Beck Depression Inventory. This inventory is a 21-item questionnaire that assesses the severity of depression. Scores can range from 0 to 63 points, with higher scores indicating a greater level of depression. Therefore, a higher score on this scale reflects a worse outcome in terms of emotional well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

REFERENCES:
- [Background] Dow B, Black K, Bremner F, Fearn M. A comparison of a hospital-based and two home-based rehabilitation programmes. Disabil Rehabil. 2007 Apr 30;29(8):635-41. doi: 10.1080/09638280600902760. PMID 17453984
- [Background] von Koch L, Wottrich AW, Holmqvist LW. Rehabilitation in the home versus the hospital: the importance of context. Disabil Rehabil. 1998 Oct;20(10):367-72. doi: 10.3109/09638289809166095. PMID 9793750
- [Background] Anderson C, Rubenach S, Mhurchu CN, Clark M, Spencer C, Winsor A. Home or hospital for stroke rehabilitation? results of a randomized controlled trial : I: health outcomes at 6 months. Stroke. 2000 May;31(5):1024-31. doi: 10.1161/01.str.31.5.1024. PMID 10797161
- [Background] Saggini R, Veraldi R, Carmignano SM, Palermo T, Russo C, Barassi G, Bellomo RG. Home Rehabilitation System in Chronic Stroke: An Observational Study in Central Italy. Neurol India. 2021 Sep-Oct;69(5):1285-1292. doi: 10.4103/0028-3886.329548. PMID 34747801
- [Background] Bickenbach J, Sabariego C, Stucki G. Beneficiaries of Rehabilitation. Arch Phys Med Rehabil. 2021 Mar;102(3):543-548. doi: 10.1016/j.apmr.2020.09.392. Epub 2020 Oct 22. PMID 33239179
- [Background] Jette AM. The Importance of Dose of a Rehabilitation Intervention. Phys Ther. 2017 Nov 1;97(11):1043. doi: 10.1093/ptj/pzx085. No abstract available. PMID 29099967
- [Background] Li G, Li X, Chen L. Personally tailored exercises for improving physical outcomes for older adults in the community: A systematic review. Arch Gerontol Geriatr. 2022 Jul-Aug;101:104707. doi: 10.1016/j.archger.2022.104707. Epub 2022 Apr 19. PMID 35462312
- [Background] Bogle Thorbahn LD, Newton RA. Use of the Berg Balance Test to predict falls in elderly persons. Phys Ther. 1996 Jun;76(6):576-83; discussion 584-5. doi: 10.1093/ptj/76.6.576. PMID 8650273
- [Background] Mat S, Tan MP, Kamaruzzaman SB, Ng CT. Physical therapies for improving balance and reducing falls risk in osteoarthritis of the knee: a systematic review. Age Ageing. 2015 Jan;44(1):16-24. doi: 10.1093/ageing/afu112. Epub 2014 Aug 22. PMID 25149678
- [Background] Hamed A, Bohm S, Mersmann F, Arampatzis A. Follow-up efficacy of physical exercise interventions on fall incidence and fall risk in healthy older adults: a systematic review and meta-analysis. Sports Med Open. 2018 Dec 13;4(1):56. doi: 10.1186/s40798-018-0170-z. PMID 30547249
- [Background] Yalew ES, Melese AZ, Guadie YG, Abich Y, Kassa T, Gashaw M. Magnitude of depression and associated risk factors among patients with musculoskeletal disorder treated in physiotherapy outpatient department in Amhara region comprehensive specialized hospital in Ethiopia: a prospective cross-sectional study. BMC Psychiatry. 2023 Mar 22;23(1):189. doi: 10.1186/s12888-023-04658-3. PMID 36949431
- [Background] Bruijniks SJ, Bosmans J, Peeters FP, Hollon SD, van Oppen P, van den Boogaard M, Dingemanse P, Cuijpers P, Arntz A, Franx G, Huibers MJ. Frequency and change mechanisms of psychotherapy among depressed patients: study protocol for a multicenter randomized trial comparing twice-weekly versus once-weekly sessions of CBT and IPT. BMC Psychiatry. 2015 Jun 30;15:137. doi: 10.1186/s12888-015-0532-8. PMID 26122891
- [Derived] Barria P, Andrade A, Gomez-Vargas D, Yelincic A, Roberti F, Bahamonde E, Aguilar R, Cordova B. Multidisciplinary Home-Based Rehabilitation Program for Individuals With Disabilities: Longitudinal Observational Study. JMIR Rehabil Assist Technol. 2024 Oct 16;11:e59915. doi: 10.2196/59915. PMID 39412860